CLINICAL TRIAL: NCT05072210
Title: Could Mobile-based Interventions Aid To "Understand and Flatten the Curve" of Stress, Anxiety, Distress and Depression Among Healthcare Providers at Unity Health Toronto During and After the COVID-19 Pandemic?
Brief Title: Mobile Interventions for the Prevention and Detection of Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Toronto Metropolitan University (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20-176; SMH-20-037 (Other Grant/Funding Number: St. Michael's Hospital AFP Innovation Fund); ML42588 (Other Grant/Funding Number: Roche Canada COVID-19 Innovation Challenge)
Record Dates: First submitted 2021-08-24; First posted 2021-10-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Depression; Anxiety; Stress; Loneliness
Keywords: Depression; Anxiety; Stress; Loneliness; Mobile Intervention
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Upon logging into the study platform, half of the participants will be automatically randomized to receive (for 4 weeks) daily-personalized automated alerts (The mobile intervention). This feature will be made available to all participants after 4 weeks. Hence, for the first 4 weeks, this study can be described as having a parallel group study model. After 4 weeks, the study switches to a single group study model, and can therefore be described as having a single group interventional model after 4 weeks from the start date until the rest of the duration of the study.
Who Masked: Participant, Investigator
Masking Description: Participants will be issued a specific ID number to be used within the mobile app to ensure that any identifiable information within this app will remain anonymous. A master linking log will serve as the only link between participants and the study data collected in the mobile app.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Intervention Group (Experimental): One half of the participants will receive personalized automated alerts throughout their involvement.
  Interventions: Other: Mobile Intervention
- Control Group (No Intervention): For 4 weeks, the other half of the participants will not receive personalized automated alerts. After 4 weeks, these alerts will be enabled.

INTERVENTIONS:
Other: Mobile Intervention — Active mobile data will be used to provide automated, personalized notifications to frontline healthcare workers. Key information on mental health and links to access additional health resources will be available on the mobile platform.
  Arms: Mobile Intervention Group

SUMMARY:
Stress, anxiety, distress and depression are exceptionally high among healthcare providers at the frontline of the COVID-19 pandemic. Knowledge of factors underlying distress and resilience and evidence based interventions to impact the mental wellbeing of frontline healthcare providers is limited. This study will evaluate a novel mobile platform to gather the "distress experience" of healthcare workers at Unity Health Toronto in real time during and after the COVID-19 pandemic, use automated personalized mobile interventions (e.g. routine, sleep, exercise) to nudge active/passive parameters to manage distress.

ELIGIBILITY:
Inclusion Criteria:

* Staff or healthcare providers working at Unity Health Toronto
* 18 years of age or older
* Must own a mobile phone running Android Version 6.0 and higher, or an iPhone 6 running OS 14 and higher)

Exclusion Criteria:

* Non-Unity Health Toronto staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | At 4 weeks from baseline
  The primary outcome measure will be the ten-item Perceived Stress Scale. Scores range from 0 to 40, and higher scores indicate more severe stress.

SECONDARY OUTCOMES:
Perceived Stress Scale | At 12 weeks from baseline
  The primary outcome measure will be the ten-item Perceived Stress Scale. Scores range from 0 to 40, and higher scores indicate more severe stress.
Active Data - Short UCLA Loneliness Scale | At 4 weeks from baseline
  Short, 3-item scale; scores range from 3 to 9, and higher scores indicate more severe loneliness symptoms. Feasibility of the mobile platform will be indicated by a significant reduction in score.
Active Data - Generalized Anxiety Disorder Scale | At 4 weeks from baseline
  7-item scale; scores range from 0 to 21, and higher scores indicate more severe anxiety symptoms. Feasibility of the mobile platform will be indicated by a significant reduction in score.
Active Data - Patient Health Questionnaire | At 4 weeks from baseline
  9-item scale; scores range from 0 to 27, and higher scores indicate more severe depression symptoms. Feasibility of the mobile platform will be indicated by a significant reduction in score.
Passive Data - GPS Sample Point Metrics | At 4 weeks from baseline
  Feasibility of the mobile platform will be determined by the number of GPS sample points (mobility metrics) collected per user per day.

CONTACTS AND LOCATIONS:
Overall Officials: Venkat Bhat, MD MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No